CLINICAL TRIAL: NCT02874261
Title: Effects of Whole Body Periodic Acceleration on Activity and Sleep In Parkinson's Disease
Brief Title: Whole Body Periodic Acceleration on Activity and Sleep In Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1124
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Sleep Disorders; Physical Activity
MeSH Terms: conditions — Sleep Wake Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole Body Periodic Acceleration (Experimental): Whole-body periodic acceleration (WBPA) is a new, non-invasive, and promising therapy for a diverse and growing list of disorders including cardiovascular disease 6. During WBPA, patients lie in the supine position on a bed that is capable of translating back and forth parallel to the ground, along the head-to-foot axis of the patient. Thus, this treatment is best described as a form of "passive exercise." The frequency of the translation is 120 cycles/minute; cpm) as well as a distance traveled 16 mm.
  Interventions: Device: Whole Body Periodic Acceleration

INTERVENTIONS:
Device: Whole Body Periodic Acceleration — oscillating bed that the subject will lie on 3 days a week for 45 minutes at 140 cycles per minute.
  Other Names: WBPA

SUMMARY:
Whole-body periodic acceleration (WBPA) is a new, non-invasive, and promising therapy for a diverse and growing list of disorders including cardiovascular disease. During WBPA, patients lie in the supine position on a bed that is capable of translating back and forth parallel to the ground, along the head-to-foot axis of the patient. Thus, this treatment is best described as a form of "passive exercise." The frequency of the translation (up to 180 cycles/minute; cpm) as well as the distance traveled (2-24mm) by the bed can be adjusted by the patient or health care professional.

The science behind the therapeutic effects of WBPA still remains largely unknown.

The investigators are observing how WBPA may impact on sleep and activity in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Sleep disturbances are common in individuals with Parkinson's Disease. Whole-body periodic acceleration (WBPA) is a new, non-invasive, and promising therapy for a diverse and growing list of disorders. During WBPA, patients lie in the supine position on a bed that is capable of translating back and forth parallel to the ground, along the head-to-foot axis of the patient. Thus, this treatment is best described as a form of "passive exercise." WBPA has been shown in previous studies to increase nitric oxide. Increased levels of nitric oxide have been shown to improve sleep patterns in other populations. The current pilot study will investigate how WBPA will impact upon sleep disturbances in subjects with Parkinson's disease who suffer from abnormal sleep patterns. The investigators will record sleep patterns and activity levels using a Jawbone U3® activity monitor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 50-80
* Individuals with Parkinsons disease between the ages of 50-80
* Individuals with a smart phone

Exclusion Criteria:

* Any condition that prevents you from lying flat on your back, any other neurological condition than Parkinson's disease.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sleep patterns using an activity monitor on the wrist | 6 weeks
  The investigators will record sleep patterns a week before WBPA through out the 4 weeks of WBPA and then one week post WBPA using an activity monitor on the wrist

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 6 weeks
  This is a quantitative tool to measure sleep as well as an activity monitor twenty -four hours for seven days at a time
Physical Activity (steps per day using an activity monitor on the wrist) | 6 weeks
  The investigators will record steps per day a week before WBPA through out the 4 weeks of WBPA and then one week post WBPA using an activity monitor on the wrist

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Southard, DPT, Principal Investigator — NYIT
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No